CLINICAL TRIAL: NCT02566304
Title: A Two Step Approach to Non-Myeloablative Allogeneic Hematopoietic Stem Cell Transplantation for Patients With Hematologic Malignancies
Brief Title: Reduced Intensity Chemotherapy and Radiation Therapy Before Donor Stem Cell Transplant in Treating Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15D.323; 2015-054 (Other: PRC); NCI-2015-01506 (Other: NCI Trial ID); JT 7773 (Other: JeffTrial Number)
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Results first posted 2025-03-20 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia in Remission; Aplastic Anemia; Chronic Myelomonocytic Leukemia; Hodgkin Lymphoma; Indolent Non-Hodgkin Lymphoma; Malignant Neoplasm; Myelodysplastic Syndrome; Myeloproliferative Neoplasm; Plasma Cell Myeloma; Refractory Anemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Ring Sideroblasts; Refractory Cytopenia With Multilineage Dysplasia; Refractory Cytopenia With Multilineage Dysplasia and Ring Sideroblasts
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Aplastic; Leukemia, Myelomonocytic, Chronic; Hodgkin Disease; Neoplasms; Myelodysplastic Syndromes; Myeloproliferative Disorders; Multiple Myeloma; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts | interventions — fludarabine; fludarabine phosphate; Whole-Body Irradiation; Cyclophosphamide; Peripheral Blood Stem Cell Transplantation; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RIC HSCT, GVHD prophylaxis (Experimental): RIC: Patients receive fludarabine phosphate IV on days -10 to -8 and cyclophosphamide IV on days -3 and -2. Patients also undergo TBI followed by a DLI on day -6.
  TRANSPLANT: Patients undergo CD34+ peripheral blood stem cell transplant on day 0.
  GVHD PROPHYLAXIS: Patients receive tacrolimus PO beginning day -1 with a taper initiated on day 42 and mycophenolate mofetil IV BID on days -1 to 28 in the absence of GVHD.
  Interventions: Drug: Fludarabine; Radiation: Total-Body Irradiation; Biological: T Cell-Depleted Donor Lymphocyte Infusion; Drug: Cyclophosphamide; Procedure: Peripheral Blood Stem Cell Transplantation; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Fludarabine — Given IV
  Other Names: Fludarabine phosphate; Fludara
Radiation: Total-Body Irradiation — Undergo TBI
Biological: T Cell-Depleted Donor Lymphocyte Infusion — Undergo DLI
Drug: Cyclophosphamide — Given IV
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune; Cycloblastin; Cytophosphane; CP
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo PBSC transplant
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo PBSC transplant
Drug: Tacrolimus — Given PO
  Other Names: FK-506; Fujimycin; Prograf; Advograf; Protopic
Drug: Mycophenolate mofetil — Given IV
  Other Names: Mycophenolic acid; MMF; CellCept; Myfortic
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This clinical trial studies the use of reduced intensity chemotherapy and radiation therapy before donor stem cell transplant in treating patients with hematologic malignancies. Giving low doses of chemotherapy, such as cyclophosphamide and fludarabine phosphate, before a donor stem cell transplant may help stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Reducing the intensity of the chemotherapy and radiation may also reduce the side effects of the donor stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate efficacy of this approach over the historical 2 step reduced intensity conditioning (RIC) approaches in the "vulnerable" population defined as: patients with hematopoietic cell transplant (HCT)-co-morbidity index (CI)/age scores >= 2, but no more than a score of 5 as based on the Sorror et al. data.

SECONDARY OBJECTIVES:

I. To compare the non-relapse mortality (NRM) and relapse related mortality (RRM) rates at 1 year for patients treated on this study to the that of patients undergoing haploidentical RIC hematopoietic stem cell transplantation (HSCT) as reported in the literature and as observed in the 2 step RIC trials.

II. To determine the incidence and severity of graft-versus-host disease (GVHD) in patients undergoing treated on the Thomas Jefferson University (TJU) RIC 2 step approach.

III. To evaluate engraftment rates and lymphoid reconstitution in patients treated on the TJU RIC 2 step approach.

OUTLINE:

RIC: Patients receive fludarabine phosphate intravenously (IV) over 60 minutes on days -10 to -8 and cyclophosphamide IV over 2 hours on days -3 and -2. Patients also undergo total body irradiation (TBI) followed by a donor lymphocyte infusion (DLI) on day -6.

TRANSPLANT: Patients undergo cluster of differentiation (CD)34+ peripheral blood stem cell transplant on day 0.

GVHD PROPHYLAXIS: Patients receive tacrolimus orally (PO) beginning day -1 with a taper initiated on day 42 and mycophenolate mofetil IV twice daily (BID) on days -1 to 28 in the absence of GVHD.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated on this study will have:

  * Acute myeloid leukemia in morphologic complete remission (CR) not requiring treatment for their disease for 4 weeks
  * A history of acute myeloid leukemia (AML) with < 10% residual blasts (use highest count on staging studies) after induction therapy and persisting with < 10% blasts for at least 8 weeks without reinduction and at the time of HSCT
  * Refractory anemia (RA) or refractory anemia with ring sideroblasts (RARS) or isolated 5q-
  * Refractory anemia with excess blasts (RAEB)-1, refractory cytopenia with multilineage dysplasia (RCMD)+/-ringed sideroblasts (RS), or myelodysplastic syndrome (MDS) not otherwise specified (NOS) with stable disease for at least 3 months
  * RAEB-2 must demonstrate chemo-responsiveness; chemo-responsiveness is defined as a persistent blast percentage decrease by at least 5 percentage points to therapy and there must be =< 10% blasts (use highest count on staging studies) after treatment and at the time of transplant
  * Hodgkin or Indolent non-Hodgkin's lymphoma
  * Myeloma with < 5% plasma cells in the marrow
  * Myeloproliferative disorders (excludes chronic myelomonocytic leukemia [CMML])
  * Aplastic anemia
  * A hematological or oncological disease (not listed) in which allogeneic HSCT is thought to be beneficial, and the disease is chemoresponsive
  * Patients without clear manifestation of their disease status in terms of stage and/or responsiveness should be discussed with the principal investigator (PI) and enrollment analysis should be documented in the study records
* Patients must have a related donor who is human leukocyte antigen (HLA) mismatched at 2, 3, or 4 antigens at the HLA-A; B; C; DR loci in the graft-versus-host disease (GVHD) direction; (patients with related donors who are HLA identical or are a 1-antigen mismatch may be treated on this therapeutic approach, but will have their outcomes will not be part of the statistical aims of the study); the HLA matched related category includes patients with a syngeneic donor
* Patients must have had front line therapy for their disease
* LVEF (left ventricular end diastolic function) of >= 45%
* DLCO (diffusing capacity of the lung for carbon monoxide) >= 45% of predicted corrected for hemoglobin, FEV-1 (forced expiratory volume at 1 second) >= 50% of predicted
* Serum bilirubin =< 1.8
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 2.5 X upper limit of normal
* Creatinine clearance of >= 60 mL/min
* HCT-CI/age score =< 5 points (patients with greater than 5 points will be allowed for trial with approval of the PI and the co-PI or his designee; this is an adjustment to account for healthy patients who meet the spirit of this protocol but have histories that result in higher than HCT-CI 5 points; an example is a patient with a solid tumor malignancy in their remote history [adds 3 points to HCT-CI total] where the treatment for the malignancy occurred years to decades before and there has been complete recovery of toxicities)
* Karnofsky performance status (KPS) >= 90% patients older than 70 years, KPS >= 80% patients younger than 70 years
* Patients must be willing to use contraception if they have childbearing potential

Exclusion Criteria:

* Performance status < 90% in patients 70 years old or greater, < 80% in patients less than age 70 years
* HCT-CI/age score > 5 points (patients with greater than 5 points will be allowed for trial with approval of the principal investigator and the co-principal investigator or his designee; this is an adjustment to account for healthy patients who meet the spirit of this protocol but have histories that result in higher than HCT-CI 5 points; an example is a patient with a solid tumor malignancy in their remote history [adds 3 points to HCT-CI total] where the treatment for the malignancy occurred years to decades before and there has been complete recovery of toxicities)
* A diagnosis of chronic myelomonocytic leukemia (CMML), unless in morphologic CR
* Human immunodeficiency virus (HIV) positive
* Active involvement of the central nervous system with malignancy
* Inability to obtain informed consent from patient or surrogate
* Pregnancy
* Patients with life expectancy of =< 6 months for reasons other than their underlying hematologic/oncologic disorder
* Patients who have received alemtuzumab or antithymocyte globulin within 8 weeks of the transplant admission; the absence of these therapies in the medical record will serve as documentation that they were not given
* Patients with evidence of another malignancy, exclusive of a skin cancer that requires only local treatment, should not be enrolled on this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Usama Gergis, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Jefferson University Hospitals — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- RIC HSCT, GVHD Prophylaxis: RIC: Patients receive fludarabine phosphate IV on days -10 to -8 and cyclophosphamide IV on days -3 and -2. Patients also undergo TBI followed by a DLI on day -6.
  TRANSPLANT: Patients undergo CD34+ peripheral blood stem cell transplant on day 0.
  GVHD PROPHYLAXIS: Patients receive tacrolimus PO beginning day -1 with a taper initiated on day 42 and mycophenolate mofetil IV BID on days -1 to 28 in the absence of GVHD.
  Fludarabine: Given IV
  Total-Body Irradiation: Undergo TBI
  T Cell-Depleted Donor Lymphocyte Infusion: Undergo DLI
  Cyclophosphamide: Given IV
  Peripheral Blood Stem Cell Transplantation: Undergo PBSC transplant
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo PBSC transplant
  Tacrolimus: Given PO
  Mycophenolate mofetil: Given IV
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | RIC HSCT, GVHD Prophylaxis
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RIC HSCT, GVHD Prophylaxis
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 24
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS will be estimated using Kaplan-Meier curves. The 1-year OS rate and corresponding 95% confidence interval will be estimated from the Kaplan-Meier curve for the OS.
Time Frame: At 1 year post HSCT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RIC HSCT, GVHD Prophylaxis
Number analyzed (Participants) | 35
percentage of participants | 74 [54 to 86]

2. Secondary Outcome: Relapse Related Mortality (RRM)
Description: Will be reported descriptively. RRM may also be estimated using Kaplan Meier curves and/or cumulative incidence analyses.
Time Frame: At 1 year post HSCT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RIC HSCT, GVHD Prophylaxis
Number analyzed (Participants) | 35
percentage of participants | 13 [4 to 28]

3. Secondary Outcome: Non-Relapse Mortality (NRM)
Description: Will be reported descriptively. NRM may also be estimated using Kaplan Meier curves and/or cumulative incidence analyses.
Time Frame: At 1 year post HSCT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RIC HSCT, GVHD Prophylaxis
Number analyzed (Participants) | 35
percentage of participants | 16 [6 to 31]

4. Secondary Outcome: Incidence and Severity of GVHD
Description: Will be reported descriptively
Time Frame: Up to 1 year post HSCT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RIC HSCT, GVHD Prophylaxis
Number analyzed (Participants) | 35
percentage of participants | 27 [13 to 43]

5. Secondary Outcome: Engraftment Rates
Description: Will be reported descriptively
Time Frame: Up to 1 year post HSCT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RIC HSCT, GVHD Prophylaxis
Number analyzed (Participants) | 35
percentage of participants | 97 [85 to 100]

6. Secondary Outcome: Lymphoid Reconstitution
Description: Lymphoid reconstitution will be evaluated monthly to every other month during the first year post HSCT and will be reported descriptively.
Time Frame: Up to 1 year post HSCT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RIC HSCT, GVHD Prophylaxis
Number analyzed (Participants) | 35
percentage of participants | 10 [3 to 25]

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed from enrollment until d+100 after transplant. All-Cause Mortality monitored/assessed up to 1 year post transplant
Description: CTCAE
Arm/Group | RIC HSCT, GVHD Prophylaxis
All-Cause Mortality (participants affected / at risk) | 1/35
Serious Adverse Events (participants affected / at risk) | 10/35
Other Adverse Events (participants affected / at risk) | 33/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIC HSCT, GVHD Prophylaxis (N=35)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) — Grade 3 - subject 3
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) — subject 33
ALT increased (Investigations) | 1 (1) — subject 13
Bilirubin increased (Investigations) | 1 (1) — subject 33
Cardiac Arrest (Cardiac disorders) | 1 (1) — subject 25
Cellulitis (Infections and infestations) | 1 (1) — subject 12
Cholecystitis (Gastrointestinal disorders) | 1 (1) — subject 3
Cognitive disturbance (Psychiatric disorders) | 2 (2) — subject 22 and subject 28
Deliurm (Psychiatric disorders) | 1 (1) — subject 19
Depressed level of Consciousness (Psychiatric disorders) | 1 (1) — subject 25
Ejection Fraction decreased (Cardiac disorders) | 1 (1) — subject 7
Fever (Infections and infestations) | 2 (2) — subject 11 & 26
Hematuria (Renal and urinary disorders) | 1 (1) — subject 1
Hepatobiliary disorder (Hepatobiliary disorders) | 1 (1) — subject 1
Hypotension (Vascular disorders) | 2 (4) — subject 25 and 28
hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 (15) — subject 1,6,7,8,12,13,25,28,33,35
Infection & Infestations- Other fever (Infections and infestations) | 1 (1) — subject 3
Lung Infection (Hepatobiliary disorders) | 2 (2)
Nervous System disorder- Aphasia (Nervous system disorders) | 1 (1) — subject 12
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — subject 12
Sepsis (Infections and infestations) | 2 (2) — subject 25 and 28
SVT (Cardiac disorders) | 1 (1) — subject 33
Syncope (General disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) — subject 10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIC HSCT, GVHD Prophylaxis (N=35)
Wound-top of head (Injury, poisoning and procedural complications) | 1 (1) — Grade 1
Wound of Groin (Injury, poisoning and procedural complications) | 1 (1) — Grade 1
Wound on buttock (Injury, poisoning and procedural complications) | 1 (1) — grade 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 (6) — grade 1
Weight loss (Metabolism and nutrition disorders) | 4 (4)
Weakness (General disorders) | 2 (2)
VRE (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 18 (31)
Volume overload (Cardiac disorders) | 3 (3) — grade 1 & 2
Vaginal cysts (Skin and subcutaneous tissue disorders) | 1 (1)
UTI-VRE (Renal and urinary disorders) | 1 (2) — grade 1
Urine incontinence (Renal and urinary disorders) | 9 (13) — grade 1
urinary retention (Renal and urinary disorders) | 8 (9) — grade 2
Urinary frequency (Renal and urinary disorders) | 12 (14) — grade 1
Trouble sleeping (Psychiatric disorders) | 1 (1) — grade 1
tooth pain (General disorders) | 2 (2) — grade 1
Tachycardia (Cardiac disorders) | 7 (11) — grade 1
Tachypnea (Cardiac disorders) | 5 (5) — grade 1
Stiff neck (Musculoskeletal and connective tissue disorders) | 1 (1) — grade 1
Sleep apnea (Psychiatric disorders) | 2 (3) — grade 2
Tinea Cruis (Infections and infestations) | 1 (1) — grade 2
Tinnitus (Ear and labyrinth disorders) | 4 (4) — grade 1
Vision changes (Eye disorders) | 1 (1) — grade 1
Urinary tract pain (Renal and urinary disorders) | 2 (2) — grade 1
Urinary Tract Infection (Renal and urinary disorders) | 6 (6) — grades 1,2,3
Typhlitis (Infections and infestations) | 1 (1) — grade 1
Vitamin K deficiency (Investigations) | 1 (1) — grade 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) — grade 2
Trouble swallowing (Gastrointestinal disorders) | 1 (1) — grade 1
Unexpected weight change (General disorders) | 1 (1) — grade 1
Tremor (Nervous system disorders) | 6 (6) — grade 1-2
Thromboembolic event (Vascular disorders) | 3 (3) — grade 1
Thrush (Infections and infestations) | 1 (1) — grade 2
Throat pain (General disorders) | 1 (1) — grade 1
sleep apnea (Psychiatric disorders) | 3 (3) — grade 2
Supraventricular tachycardia (Cardiac disorders) | 2 (2) — grade 2
tissue disorders- other, skin tear (Skin and subcutaneous tissue disorders) | 1 (1) — grade 1
Skin and Subcutaneous tissue disorders-other, sacrum sore (Skin and subcutaneous tissue disorders) | 1 (1) — grade 2
Skin and subcutaneous tissue disorders- other, erythema (Skin and subcutaneous tissue disorders) | 3 (3) — grade 1
Skin and subcutaneous tissue disorders- other, keratosis (Skin and subcutaneous tissue disorders) | 1 (1) — grade 2
skin and subcutaneous tissue disorders- other, Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) — grade 1
Skin and subcutaneous tissue disorders, other excoriation (Skin and subcutaneous tissue disorders) | 1 (1) — grade 2
Syncope (General disorders) | 2 (2) — grade 3
Somnolence (Psychiatric disorders) | 2 (2) — grade 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) — grade 1
Skin- Ashen color (Skin and subcutaneous tissue disorders) | 1 (1) — grade 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) — grade 1-
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — grade 1
sinus tachycardia (Cardiac disorders) | 17 (30) — grade 1-2
Sinus Bradycardia (Cardiac disorders) | 1 (1) — grade 3
Shoulder pain (Musculoskeletal and connective tissue disorders) | 3 (3) — grade 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 4 (4) — grade 1
Sexual dysfunction (Vascular disorders) | 1 (1) — grade 1
sore throat (Gastrointestinal disorders) | 2 (2) — grade 1
Skin peeling (Skin and subcutaneous tissue disorders) | 2 (3) — grade 1
subconjunctiva hemorrhage (Eye disorders) | 1 (1) — grade 1
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) — grade 1
scalp pain (General disorders) | 1 (1) — grade 1
Scrotal pain (Reproductive system and breast disorders) | 3 (3) — grade 1
Scrotal Edema (Reproductive system and breast disorders) | 2 (2) — grade 2
scleral disorder (Skin and subcutaneous tissue disorders) | 1 (1) — grade 1
Sepsis (Infections and infestations) | 1 (1) — grade 4
Right arm swelling (Cardiac disorders) | 1 (1) — grade 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — grade 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — grade 1
Rash (Skin and subcutaneous tissue disorders) | 17 (23) — grade 1-2
Respiratory, thoracic and mediastinal disorders- other, rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) — grade 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 (19) — grade 1-3
Rigors (General disorders) | 1 (2) — grade 1
Renal and urinary disorders- other, dysuria (Renal and urinary disorders) | 2 (2) — grade 1
Rectal pain (General disorders) | 4 (4) — grade 1
Respiratory, thoracic and mediastinal disorders- other, nasopharyngeal bleed (Respiratory, thoracic and mediastinal disorders) | 1 (1) — grade 1
Renal and Urinary disorders- hemorrhagic cystitis due to BK virus (Renal and urinary disorders) | 1 (1) — grade 3
Reproductive system and breast disorders- other, scrotal edema (Reproductive system and breast disorders) | 1 (1) — grade 2
Renal and urinary disorders- other, decreased urine output (Renal and urinary disorders) | 10 (12) — grade 1-2
Respiratory, thoracic and mediastinal disorders - other, tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — grade 2
Renal and Urinary disorders- other, difficulty urinating (Renal and urinary disorders) | 1 (1) — grade 1
Premature Ventricular Contractions (Cardiac disorders) | 1 (1) — grade 2
Pulmonary edema (Cardiac disorders) | 3 (3) — grade 1
Pruritis (Skin and subcutaneous tissue disorders) | 10 (11) — grade 1-2
Pleural effusions (Respiratory, thoracic and mediastinal disorders) | 4 (4) — grade
Pericardial effusion (Cardiac disorders) | 6 (6) — grade 1-2
Vasovagal reaction (Nervous system disorders) | 1 (1) — grade 3
Skin and subcutaneous tissue disorders- other, diaphoretic (Skin and subcutaneous tissue disorders) | 1 (1) — grade 2
Skin and subcutaneous disorders- other, pale (Skin and subcutaneous tissue disorders) | 1 (1) — grade 1
viral conjunctivitis (Eye disorders) | 1 (1) — grade 1
Unspecified eye problem (Eye disorders) | 1 (1) — grade 1
taste change (General disorders) | 1 (1) — grade 1
sleep disturbance (Psychiatric disorders) | 2 (2) — grade 1
skin and subcutaneous tissue disorders- other, Pallor (Skin and subcutaneous tissue disorders) | 1 (1) — grade 1
sinus headache (Nervous system disorders) | 1 (1) — grade 1
Paresthesia pain (Nervous system disorders) | 4 (4) — grade 1
Palpitations (Cardiac disorders) | 2 (4) — grade 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (16) — grades 1-2
Pain - general (General disorders) | 10 (12) — grades 1-2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — grade 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (4) — grade 1-2
Pneumonitis (Infections and infestations) | 1 (1) — grade 3
Parotiditis (Infections and infestations) | 3 (3) — grade 1
Physical deconditioning (General disorders) | 2 (2) — grade 2
Psychiatric disorders- other, decreased concentration (Psychiatric disorders) | 3 (3) — grade 1
Pericarditis (Cardiac disorders) | 1 (1) — grade 2
Peripheral neuropathy (Nervous system disorders) | 4 (4) — grade 1
peripheral edema (General disorders) | 2 (2) — grade 1-2
patchy spots on tongue (Skin and subcutaneous tissue disorders) | 1 (1) — grade 2
Pruritic raised erythematous rash (Skin and subcutaneous tissue disorders) | 1 (1) — grade 2
polyuria (Renal and urinary disorders) | 1 (1) — grade 1
Odynophagia (Gastrointestinal disorders) | 1 (1) — grade 1
Night sweats (Blood and lymphatic system disorders) | 3 (3) — grade 1
Neuro-weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — grade 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 (5) — grade 1
Nausea (Gastrointestinal disorders) | 20 (31) — grade 1-2
Non- cardiac chest pain (General disorders) | 3 (3) — grade 1
Nervous System Disorders- other, Altered MS with Aphasia (Nervous system disorders) | 1 (1) — grade 3
Neoplasms benign, malignant and unspecified (in cyss and polyps)- other, bump on left arm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — grade 1
Nosebleeds (General disorders) | 2 (2) — grade 1
Nocturia (Renal and urinary disorders) | 2 (2) — grade 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) — grade 1-2
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) — grade 1
Mucositis (Respiratory, thoracic and mediastinal disorders) | 21 (22) — grade 3
MRSA - skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) — grade 2
Musculoskeletal and connective tissue disorder- other, Charlie HOrse (Musculoskeletal and connective tissue disorders) | 1 (1) — grade 1
Musculoskeletal and connective tissue disorders- other, unsteadiness on feet (Musculoskeletal and connective tissue disorders) | 2 (2) — grade 2
Malaise (General disorders) | 4 (6) — grade 1-2
Memory impairment (Psychiatric disorders) | 3 (3) — grade 2
Musculoskeletal and connective tissue disorders- other, physical deconditioning (Musculoskeletal and connective tissue disorders) | 1 (1) — grade 2
Muscle weakness in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) — grade 1
Metabolism and nutrition disorders- electrolyte disturbances (Metabolism and nutrition disorders) | 1 (1) — grade 3
Mouth Sores (Gastrointestinal disorders) | 1 (1) — grade 1
Lung Infection (Hepatobiliary disorders) | 3 (3) — grade 2-3
Lump on right forearm (Endocrine disorders) | 1 (1) — grade 1
Loss of smell/taste (Nervous system disorders) | 1 (1) — grade 1
Loose Stools (Gastrointestinal disorders) | 1 (1) — grade 1
Lightheadedness (Vascular disorders) | 3 (4) — grade 1
Lethargy/Fatigue (General disorders) | 3 (4) — grade 2
Left pericatheter thrombus (Blood and lymphatic system disorders) | 1 (1) — grade 1
LE edema (General disorders) | 1 (1) — grade 1
Left Axilla swelling (Blood and lymphatic system disorders) | 1 (1) — grade 1
Itching (Skin and subcutaneous tissue disorders) | 1 (1) — grade 1
Irregular heart ryhythm (Cardiac disorders) | 1 (1) — grade 1
Insomnia (Psychiatric disorders) | 15 (19) — grade 1-2
Infusion Related Reaction - rigors (Infections and infestations) | 1 (1) — grade 2
Infusion related reaction- Hypertension (Cardiac disorders) | 1 (1) — grade 1
Infusion related reaction- headache (Nervous system disorders) | 1 (1) — grade 1-2
Infusion related reaction- chills (Infections and infestations) | 2 (2) — grade 1-2
infusion related reaction (General disorders) | 12 (13) — grade 1-2
Infection and Infestations- other (fever) (Infections and infestations) | 4 (4) — grade 3
Indigestion (Gastrointestinal disorders) | 1 (1) — grade 1
Increased LFT's (Hepatobiliary disorders) | 1 (1) — grade 1
infections and infestations- other, CMV reactivation (Infections and infestations) | 1 (1) — grade 1
Infections and infestations- other, cellulitis (Infections and infestations) | 1 (1) — grade 3
increased creatinine (Investigations) | 6 (6) — grade 1
Iron overload (Investigations) | 2 (2) — grade 1
Injury, poisoning and procedural complications- other, wounds (Injury, poisoning and procedural complications) | 2 (2) — grade 2
injury, poisoning and procedural complications- other, scrotal bleeding (Injury, poisoning and procedural complications) | 1 (1) — grade 2
injury, poisoning and procedural complications- other, pressure ulcer (Injury, poisoning and procedural complications) | 1 (1) — grade 1
injury, poisoning and procedural complications- other, parotitis (Injury, poisoning and procedural complications) | 1 (1) — grade 2
injury, poisoning and procedural complications- other, GI bleeding (Injury, poisoning and procedural complications) | 1 (1) — grade 3
Infusion related reaction- hypotension (Vascular disorders) | 1 (1) — grade 1
Infections and infestations- other, HHV-6 (Infections and infestations) | 1 (1) — grade 2
Infections and infestations- other, CMV Viremia (Infections and infestations) | 1 (1) — grade 2
Infections and infestations- other, bacteremia (Infections and infestations) | 4 (4) — grade 3
injury, poisoning and procedural complications- other ecchymosis (Injury, poisoning and procedural complications) | 1 (1) — grade 1
infections and infestations- other, epididmoorchitis (Infections and infestations) | 1 (1) — grade 3
infections and infestations- other, covid-19 (Infections and infestations) | 1 (1) — grade 1
intermittent hyperglycemia (Investigations) | 1 (1) — grade 1
intermittent headache (Nervous system disorders) | 1 (1) — grade 1
intermittent fatigue (General disorders) | 2 (2) — grade 1
intermittent dizziness (Nervous system disorders) | 1 (1) — grade 1
Vaginal Pain (Reproductive system and breast disorders) | 1 (1) — grade 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (2) — grade 2
Phantom pain (General disorders) | 1 (1) — grade 2
Oral Pain (General disorders) | 1 (1) — grade 2
Metabolism and nutritional disorders- other, vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) — grade 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 19 (25) — grade 2-3
Hypotension (Vascular disorders) | 18 (35)
Hypothyroidism (Endocrine disorders) | 1 (1) — grade 2
Hypertension (Vascular disorders) | 12 (16) — grade 1-2
Hyperkalemia (Endocrine disorders) | 7 (7) — grade 2
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) — grade 2
Hot flashes (Reproductive system and breast disorders) | 3 (3) — grade 1
Hive (Immune system disorders) | 1 (1) — grade 1
Hematuria (Renal and urinary disorders) | 14 (20) — grade 1
Headache (General disorders) | 13 (27) — grade 1-2
Hallucinations (Psychiatric disorders) | 6 (8) — grade 1
Hiccups (General disorders) | 3 (3) — grade 1-2
Hematuria (Renal and urinary disorders) | 1 (1) — grade 2
Hypomagnesemia (Investigations) | 6 (6) — grade 3
Hypokalemia (Investigations) | 6 (6) — grade 1
Hyperglycemia (Investigations) | 2 (2) — grade 3
Hypothermia (Investigations) | 3 (5) — grade 2
Hypophosphatemia (Investigations) | 1 (1) — grade 3
Hyponatremia (Investigations) | 4 (5)
Hypernatremia (Investigations) | 5 (5) — grade 3
Heel pain (General disorders) | 1 (1) — grade 1
Hyperhidrosis (General disorders) | 1 (1) — grade 1
Hoarsness (Respiratory, thoracic and mediastinal disorders) | 1 (2) — grade 1
hemorrhoids (Skin and subcutaneous tissue disorders) | 1 (1) — grade 1
Hyperphosphatemia (Investigations) | 1 (1) — grade 1
GERD (Gastrointestinal disorders) | 7 (7) — grade 1-2
General Disorders and administration site conditions - other Diaphoresis (General disorders) | 1 (2) — grade 1
General disorders and administration site conditions- other, generalized aches (General disorders) | 1 (1) — grade 1
Gastrointestinal disorders- other, Oral ulcer (Gastrointestinal disorders) | 1 (1) — grade 1
Gait Disturbance (Musculoskeletal and connective tissue disorders) | 7 (8) — grade 2
General disorders and administration site conditions- other fluid overload (General disorders) | 8 (10) — grade 2
Gatrointestinal disorders- other oral blister (Gastrointestinal disorders) | 2 (2) — grade 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (4) — grade 2
Gastrointestinal disorders- other, "itchy" mouth (Gastrointestinal disorders) | 1 (1) — grade 1
General disorders and administration site disorders- other, night sweats (General disorders) | 1 (1) — grade 1
general disorders and administration site conditions- other, bleeding event (General disorders) | 1 (1) — grade 1
gastrointestinal pain (General disorders) | 1 (1) — grade 1
gastrointestinal disorders- other, Perirectal irritation (Gastrointestinal disorders) | 1 (1) — grade 1
gastrointestinal disorders- other, pain at PEG site (Gastrointestinal disorders) | 1 (1) — grade 2
gastrointestinal disorders- other, hematochezia (Gastrointestinal disorders) | 1 (1) — grade 1
Gastrointestinal disorders- other, tongue coating (Gastrointestinal disorders) | 1 (1) — grade 1
Generalized itching (Skin and subcutaneous tissue disorders) | 1 (1) — grade 1
Hypervolemia (General disorders) | 3 (3) — grade 2
Foot and Leg pain (Musculoskeletal and connective tissue disorders) | 1 (3) — grade 1
Flatulence (Gastrointestinal disorders) | 11 (12) — grade 1
Fever (Infections and infestations) | 31 (63) — grade 1-3
Fatigue (General disorders) | 29 (34) — grade 1 -3
Fall (Injury, poisoning and procedural complications) | 4 (4) — grade 1
Flushing (General disorders) | 1 (1) — grade 1
Floaters (Eye disorders) | 1 (1) — grade 1
Epistaxis (Blood and lymphatic system disorders) | 4 (4) — grade 1
Enterocolitis (Gastrointestinal disorders) | 1 (1) — grade 2
Elevated total bilirubin level (Hepatobiliary disorders) | 1 (1) — grade 2
Elevated creatinine (Blood and lymphatic system disorders) | 1 (1) — grade 1
Ejection fraction decreased (Cardiac disorders) | 3 (3) — grade 3
Edema (Cardiac disorders) | 17 (25) — grade 1-2
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) — grade 1
Ear pain (Ear and labyrinth disorders) | 2 (2) — grade 1
Eye disorders - other, blind in right eye (Eye disorders) | 1 (1) — grade 2
Eye infection (Eye disorders) | 1 (1) — grade 2
Eye disorders, other Diplopia (Eye disorders) | 2 (2) — grade 1
Excoriation - scrotum (Reproductive system and breast disorders) | 1 (1) — grade 1
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) — grade 1
ear and labyrinth disorders- other, ear fullness (Ear and labyrinth disorders) | 1 (1) — grade 1
eye disorders- other, farsightedness (Eye disorders) | 1 (1) — grade 1
Extrapyramidal disorder (Nervous system disorders) | 1 (1) — grade 2
Esophagitis (Gastrointestinal disorders) | 1 (1) — grade 2
Dysuria (Renal and urinary disorders) | 3 (3) — grade 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 (23) — grade 1
DVT (Blood and lymphatic system disorders) | 2 (2) — grade 2
Dry mouth (Gastrointestinal disorders) | 10 (12) — grade 1
Dry Eyes (Eye disorders) | 4 (5) — grade 1-2
Double vision (Eye disorders) | 2 (2) — grade 1
Diarrhea (Gastrointestinal disorders) | 32 (59) — grade 1-2
Distended stomach (Gastrointestinal disorders) | 1 (1) — grade 1
Discomfort at foley site (Injury, poisoning and procedural complications) | 1 (1) — grade 1
Depression (Psychiatric disorders) | 11 (13) — grade 1-2
decreased PO intake (Metabolism and nutrition disorders) | 1 (1) — grade 1
decreased appetite (Metabolism and nutrition disorders) | 2 (3) — grade 1
Dyspepsia (Gastrointestinal disorders) | 2 (2) — grade 2
Dizziness (Nervous system disorders) | 10 (14) — grade 1-2
Delirium (Psychiatric disorders) | 6 (7) — grade 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) — grade 1-2
Diaphoresis (General disorders) | 1 (1) — grade 1
Dysphagia (Gastrointestinal disorders) | 5 (6) — grade 2
Dysgeusia (Gastrointestinal disorders) | 1 (1) — grade 1
Distention (Gastrointestinal disorders) | 1 (1) — grade 1
deconditioning (General disorders) | 1 (1) — grade 2
dehyrdration (General disorders) | 3 (3) — grade 1-2
cough (Respiratory, thoracic and mediastinal disorders) | 13 (18) — grade 1-2
cystitis noninfective (Renal and urinary disorders) | 2 (2) — grade 2
constipation (Gastrointestinal disorders) | 15 (20) — grade 1
Confusion (Psychiatric disorders) | 9 (14) — grade 1-2
CMV reactivation (Infections and infestations) | 1 (1) — grade 2
chills (General disorders) | 12 (16) — grade 1
chest tightness (Cardiac disorders) | 1 (1) — grade 1
chest pain (Cardiac disorders) | 5 (5) — grade 1
Cardio disorders- other, murmur (Cardiac disorders) | 1 (1) — grade 1
crushingoid (General disorders) | 1 (1) — grade 1
cognitive disturbance (Psychiatric disorders) | 4 (4) — grade 3
crackles at lung bases (Respiratory, thoracic and mediastinal disorders) | 1 (1) — grade 1
cholelithiasis (General disorders) | 1 (1) — grade 2
cytomegalovirus viremia (Infections and infestations) | 1 (1) — grade 3
burning sensation (Renal and urinary disorders) | 1 (1) — grade 1
blood bilirubin increased (Hepatobiliary disorders) | 13 (22) — grade 1-2
bladder pressure (Renal and urinary disorders) | 1 (1) — grade 1
bibasilar atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — grade 1
back pain and stiffness (Musculoskeletal and connective tissue disorders) | 12 (13)
buttocks pain (General disorders) | 1 (1) — grade 1
bruising (Skin and subcutaneous tissue disorders) | 2 (2) — grade 1
bradycardia (Cardiac disorders) | 1 (1) — grade 1
bloating (Gastrointestinal disorders) | 1 (1) — grade 1
blood and lymphatic system disorders- other (Blood and lymphatic system disorders) | 1 (1) — grade 5
bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) — grade 1
blood blister (Skin and subcutaneous tissue disorders) | 1 (1) — grade 1
bone pain (General disorders) | 1 (2) — grade 1-2
bilateral pam itching (Skin and subcutaneous tissue disorders) | 1 (1) — grade 1
bilateral leg cramp (General disorders) | 1 (1) — grade 1
bilateral edema (General disorders) | 1 (1) — grade 1
awakening to urinate (Renal and urinary disorders) | 3 (3) — grade 1
atrial fibrillation (Cardiac disorders) | 2 (5) — grade 2
asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) — grade 1
Anxiety (Psychiatric disorders) | 6 (7) — grade 1
Alopecia (Skin and subcutaneous tissue disorders) | 11 (11) — grade 1
Agitated/ Irritable (Psychiatric disorders) | 2 (2) — grade 1
Acidy mouth (Gastrointestinal disorders) | 1 (1) — grade 1
Achiness (Musculoskeletal and connective tissue disorders) | 1 (1) — grade 1
Abrasion (Gastrointestinal disorders) | 2 (2) — grade 1
Abdominal pain (Gastrointestinal disorders) | 19 (28) — grade 1-2
aspartate aminotransferase increased (Investigations) | 4 (5) — grade 1
arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) — grade 1
alkaline phosphate increased (Investigations) | 5 (6) — grade 1
abdominal distention (Gastrointestinal disorders) | 7 (8) — grade 1
anorexia (General disorders) | 20 (22) — grade 1-2
alanine aminotransferase increased (Investigations) | 4 (6) — grade 1-4
acute kidney injury (Renal and urinary disorders) | 10 (13) — grade 1-2
aspiration (Gastrointestinal disorders) | 1 (1) — grade 1
Atrial Flutter (Cardiac disorders) | 1 (1) — grade 2
ascites (Gastrointestinal disorders) | 1 (1) — grade 1
altered taste (General disorders) | 1 (1) — grade 1
atrial fibrillation RVR (Cardiac disorders) | 1 (1) — grade 1
acute diverticulitis (Gastrointestinal disorders) | 1 (1) — grade 1
abdominal discomfort (Gastrointestinal disorders) | 1 (1) — grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT02566304/Prot_SAP_000.pdf